CLINICAL TRIAL: NCT01853891
Title: Effects of Sleeping With Dim Light at Night in Patients With Obstructive Sleep Apnea
Brief Title: Dim Light at Night in Patients With Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of funding.
Sponsor: Ulysses Magalang MD (Other)
Responsible Party: Sponsor-Investigator, Ulysses Magalang MD, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2012H0315
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2016-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual condition (No Intervention): sleep in usual room light condition for 5 nights
- dLAN (Experimental): sleep with dim light at night for 5 nights
  Interventions: Other: dim light at night

INTERVENTIONS:
Other: dim light at night
  Arms: dLAN

SUMMARY:
With the advent of electricity, light at night has become a ubiquitous part of our society.

The main purpose of this study is to determine whether sleeping with dim light (40 lux), the brightness of a night light) in your bedroom for 5 consecutive nights will result in increased markers of inflammation in the blood compared to sleeping in darkness during the night in patients with obstructive sleep apnea (OSA).

A secondary aim is to examine the effects on insulin sensitivity, other blood proteins, and RNA molecules as a result of sleeping with dim light. RNA molecules are substances in blood that dictate what type of proteins the body should make.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether sleeping with dLAN (40 lux) for 5 consecutive nights will result in increased markers of inflammation compared to sleeping in darkness (< 1 lux) during the night in patients with OSA. A secondary aim is to examine the effects on insulin sensitivity, adipokines, and RNA molecules.

The risks associated with this study are minimal compared to the potential benefits. Knowledge about the effects of sleeping with dim light on inflammation in patients with OSA is important and would guide future recommendations about proper sleep hygiene. This research may also guide future recommendations about light conditions in other environments such as hospital bedrooms.

ELIGIBILITY:
Inclusion Criteria:

* • 18 -60 years of age.

  * Willing and able to give informed consent
  * AHI >10 episodes per hour based on a prior PSG.
  * Patients who have been started on treatment for OSA with either Continuous Positive Airway Pressure (CPAP) or dental device will be eligible for the study as long as they have been compliant with treatment for at least 30 days.

Exclusion Criteria:

* • Incapable of giving informed consent

  * Under the age of 18
  * Currently sleeping with lights on in the bedroom
  * Excessive alcohol consumption

    * Excessive alcohol use is defined as:
    * More than 3 glasses of wine a day
    * More than 3 beers a day
    * More than 60 mL of hard liquor a day
  * Room air oxyhemoglobin saturation < 88%
  * Use of home oxygen
  * Use of corticosteroids and other immunosuppressive medications.
  * Diagnosis of: HIV, Connective Tissue Disease (Lupus, Rheumatoid arthritis), Inflammatory Bowel Disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Exposure to Dim Light at Night | 5 consecutive nights
  The main purpose of this study is to determine whether sleeping with dim light (40 lux), the brightness of a night light) in your bedroom for 5 consecutive nights will result in increased markers of inflammation in the blood compared to sleeping in darkness during the night in patients with obstructive sleep apnea (OSA).

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalnag, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States